CLINICAL TRIAL: NCT05543980
Title: Home-based Leg Heat Therapy to Improve Walking Performance in Elderly Individuals: a Pilot Trial
Brief Title: Leg Heat Therapy in Elderly Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Indiana Clinical and Translational Sciences Institute (Other); American College of Sports Medicine Foundation (Unknown)
Responsible Party: Principal Investigator, Bruno Roseguini, Associate Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2022-381
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Aging; Muscle Weakness
Keywords: heat therapy; aging; muscle strength
MeSH Terms: conditions — Muscle Weakness; Hyperthermia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham control (Sham Comparator): Participants will be provided a leg heat therapy system and will be instructed to apply the therapy daily (90 min/day) for 12 consecutive weeks. The water heater will circulate water at 33ºC.
  Interventions: Device: Sham device
- Heat therapy (Experimental): Participants will be provided a leg heat therapy system and will be instructed to apply the therapy daily (90 min/day) for 12 consecutive weeks. The water heater will circulate water at 42ºC.
  Interventions: Device: Leg heat therapy device

INTERVENTIONS:
Device: Sham device — The leg heat therapy device consists of a water tank coupled with a circulator, a sous-vide water heater and water-circulating trousers. The water heater in the sham device is adjusted to heat up the water to 33ºC.
  Arms: Sham control
Device: Leg heat therapy device — The leg heat therapy device consists of a water tank coupled with a circulator, a sous-vide water heater and water-circulating trousers. The water heater in the sham device is adjusted to heat up the water to 42ºC.
  Arms: Heat therapy

SUMMARY:
This pilot randomized, sham-controlled trial aimed to establish the feasibility and safety of home-based leg HT in community-dwelling older adults and inform the design of a future, larger study. Participants were randomized to either an HT or a sham group and were asked to apply the treatment daily for 90 min over 12 consecutive weeks. The primary outcomes were compliance with the HT regimen, measured by a hidden timer, completion rates, and device safety. The secondary goals were to examine the effects of leg HT on 6-min walk distance, sit-to-stand performance, blood pressure, quality of life, and the morphology and strength of the calf muscles, as assessed using combined T1-weighted and mDixon magnetic resonance imaging (MRI). Building upon previous findings in young individuals, preclinical models of PAD, and older individuals with PAD, we hypothesized that older adults treated with leg HT for 12 weeks would display improved walking performance, increased calf strength, and reduced intramuscular fat when compared to sham-treated individuals.

DETAILED DESCRIPTION:
Aging and a sedentary lifestyle are associated with a progressive deterioration of skeletal muscle contractile function and cardiorespiratory fitness, resulting in an impaired capacity to perform daily activities and maintain independent functioning. Few therapeutic options exist to combat the skeletal muscle abnormalities and restore muscle strength in older individuals. Heat therapy (HT) is a practical, non-invasive therapeutic tool that has been shown to elicit beneficial adaptations in both vasculature and skeletal muscle. This pilot randomized, sham-controlled trial aimed to establish the feasibility and safety of home-based leg HT in community-dwelling older adults and inform the design of a future, larger study. Participants were randomized to either an HT or a sham group and were asked to apply the treatment daily for 90 min over 12 consecutive weeks. The primary outcomes were compliance with the HT regimen, measured by a hidden timer, completion rates, and device safety. The secondary goals were to examine the effects of leg HT on 6-min walk distance, sit-to-stand performance, blood pressure, quality of life, and the morphology and strength of the calf muscles, as assessed using combined T1-weighted and mDixon magnetic resonance imaging (MRI). Building upon previous findings in young individuals, preclinical models of PAD, and older individuals with PAD, we hypothesized that older adults treated with leg HT for 12 weeks would display improved walking performance, increased calf strength, and reduced intramuscular fat when compared to sham-treated individuals.

ELIGIBILITY:
Participants must be:

1. 65 yrs or older
2. Sedentary - Exercise less than three days/week, 20 minutes per day.
3. Non smokers

The exclusion criteria consisted of:

1. smoking
2. reliance on a walking aid other than a cane
3. having active cancer
4. inability to fit into water-circulating trousers
5. inability to complete the 6-minute walk test
6. being under 65 years of age
7. scoring less than 23 on the Mini-Mental Status Examination (MSSE)
8. having impaired thermal sensation in the leg

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Compliance | Baseline to 12-week follow-up
  A built-in timer inside the pump that is inaccessible to participants will provide one assessment of patient compliance with the therapy. Compliance will be determined by dividing the number of hours of HT recorded use by the required hours. In addition, patients in both groups will receive a logbook to record their treatment sessions.
Completion rate | Baseline to 12-week follow-up
  Completion rates will be defined as the number of patients attending the follow-up assessments.
Safety | Baseline through 12-week follow-up
  The study coordinator will call patients weekly to record: 1) the dates and times in which the treatment was applied, 2) BP values prior to and immediately after the end of each session, 3) the occurrence of symptoms, such as faintness or dizziness after exposure to the therapy, and 4) changes in medical status or medications. Adverse events (AEs) will be tracked throughout the study and used as a surrogate for safety-related outcomes.

SECONDARY OUTCOMES:
Triceps surae peak torque | Baseline to 12-week follow-up
  The investigators will determine whether home-based leg heat therapy improves the peak torque of the triceps surae at 12-week follow-up compared to the sham treatment.
Repeated chair rises | Baseline to 12-week follow-up
  The investigators will determine whether home-based leg heat therapy improves the time to complete 5 chair rises at 12-week follow-up compared to the sham treatment.
Short-Form (SF)-36 Questionnaire | Baseline to 12-week follow-up
  The investigators will determine whether home-based leg heat therapy improves the score in the Short-Form (SF)-36 Questionnaire at 12-week follow-up compared to the sham treatment.
Triceps sure volume and cross-sectional area | Baseline to 12-week follow-up
  The investigators will determine whether home-based leg heat therapy enhances the volume and cross-sectional area of the triceps sure at 12-week follow-up compared to the sham treatment.
Triceps sure fat content | Baseline to 12-week follow-up
  The investigators will determine whether home-based leg heat therapy reduces the fat content of the triceps sure at 12-week follow-up compared to the sham treatment.
Six-minute walk distance | Baseline to 12-week follow-up
  The investigators will determine whether home-based leg heat therapy improves the 6-minute walk distance at 12-week follow-up compared to the sham treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States